CLINICAL TRIAL: NCT07025694
Title: Feasibility Testing of a Homebased Exercise Intervention in Children With Cerebral Palsy Who Are Ambulant - The HOME-EX Study
Brief Title: Exercise Training Among Children With Cerebral Palsy to Increase Health and Well-being - A Feasibility Study
Acronym: HOME-EX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Åsa Tornberg, Associate Professor and Senior LEcturer, Lund University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LU_HOME-EX2025
Record Dates: First submitted 2025-04-23; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Children With Cerebral Palsy Who Are Ambulant; Cerebral Palsy GMFCS-ER I-II
Keywords: Children; Cerebral Palsy; Exercise; Feasibility; MICT; HIIT; eHealth; Home based exercise
MeSH Terms: conditions — Cerebral Palsy; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Children with Cerebral Plasy who are Ambulant (CP-A) (Other): Children with CP-A defined classified with the 5-level Gross Motor Function Classification System Expanded & Revised (as GMFCS-E&R) as GMFCS-E&R I-II.
  Interventions: Device: A eHealth application on a computer tablet contected to a secure severer with an interface on a computer to deliver exercise interventions.; Device: A eHealth application on a computer tablet contected to a secure severer with an interface on a computer to deliver exercise interventions; Other: Moderate Intensity Continues Training; Other: High intensity interval training
- Children who are Typically Developted (TD) (Other): Ambulant children who are TD with no other neurological diagnoses, metabolic diagnoses, orthopaedic disabilities, asthma, heart diseases, cognitive impairment, or indigestion of regular medication.
  Interventions: Device: A eHealth application on a computer tablet contected to a secure severer with an interface on a computer to deliver exercise interventions.; Device: A eHealth application on a computer tablet contected to a secure severer with an interface on a computer to deliver exercise interventions; Other: Moderate Intensity Continues Training; Other: High intensity interval training

INTERVENTIONS:
Device: A eHealth application on a computer tablet contected to a secure severer with an interface on a computer to deliver exercise interventions. — Feasibility, acceptability and usability testing of delivering home-based exercise MICT and HIIT via a Vidoe-call at fixed time-points. Tuesday, Thursday, Saturday during the 3 week-period of supervision via zoom.
  Other Names: Vidoecall exercise
Device: A eHealth application on a computer tablet contected to a secure severer with an interface on a computer to deliver exercise interventions — Feasibility, acceptability and usability testing of delivering home-based exercise MICT and HIIT via a pre-recorded videos at convenient time-point with at least one day in between during the periods of video-supervision
  Other Names: Pre-recorded exercise
Other: Moderate Intensity Continues Training — The MICT exercise training on a spinning-bike will consist of moderate intensity-longer (60%Wpeak) duration exercise carried out 3 times per week. Tuesday, Thursday, Saturday during the 3 week-period of supervision via zoom, and at time-point with at least one day in between during the periods of video-supervision. Exercise will consist of continuous biking at an individualized workload based on pre-exercise testing, for a total time of 30 minutes.
  Other Names: MICT
Other: High intensity interval training — The HIIT exercise training on a spinning-bike will begin by using a protocol consisting of bouts of high-intensity (95%Wpeak) exercise lasting for 60 seconds. These bouts will be interspersed by 4 minutes of low intensity exercising (40%Wpeak). There will be 5 bouts per session. Exercise will consist of continuous biking at individualized workloads based on pre-exercise testing. The exercise will be carried out 3 times per week. Tuesday, Thursday, Saturday during the 3 week-period of supervision via zoom, and at time-point with at least one day in between during the periods of video-supervision.
  Other Names: HIIT

SUMMARY:
The use of eHealth in children with cerebral palsy (CP) holds promise to increase participation in exercise. eHealth, has shown to increase accessibility to appropriate healthcare professionals as well as reduces time- and energy consuming transportation to/from physical appointments[5]. In children with CP reduced transportation to and from appointments, increased access to appropriate healthcare s professionals have shown to increase exercise.

However, the knowledge on how eHealth can support children with CP to participate in exercise is scarce and to the best of our knowledge there are no studies studying eHealth to increase exercise in children with CP. If HOME-EX research project is successful, we will unravel knowledge that will facilitate implementation of prescription of targeted, personalized exercise regimes to children with CP to enhance health and wellbeing and furthermore set a healthy lifestyle.

PURPOSE AND AIMS

The overall goal of the HOME-EX project is to develop, feasibility test, pilot the efficacy and map the conditions for future implement an eHealth application to support participation in exercise at home in children with CP who are ambulant (CP-A). The specific aims are:

Aim 1: From a pre-exciting eHealth-solution develop an application for Android-based tablet supporting exercise in the home of the children with CP-A in co-creation with children, family caregivers, professional caregivers, sports professionals and researchers.

Aim 2: Develop exercise sessions, as online supervised session and pre-video recorded sessions in co-creation with children, family caregivers, professional caregivers, sports professionals and researchers, to be delivered by the eHealth-solution.

Aim 3: To study the feasibility of the delivery of the exercise sessions from the eHealth-solution.

PROJECT DESCRIPTION Cerebral palsy (CP) is the most common physical disability in childhood, approximately 1.6/1000 children have CP with affected muscle tone, movement and motor skills, often accompanied by pain, epilepsy and intellectual, communicational and behavioural impairment.

The degree of motor impairment in CP is extremely variable and classified with the 5-level Gross Motor Function Classification System Expanded & Revised (GMFCS-E&R). Children with CP-A (GMFCS-E&R level I-II) can either walk and/ stand independently.

Project management Since children are non-autonomous, the common point of departure for our research is the family; lifestyle changes as well as interventions must be implemented through the family. Feasibility testing aims to analyse clinical, procedural, and methodological uncertainties of the exercise testing and the exercise training interventions designed in co-creation with stakeholders. If no major changes are made to the study design and/or the intervention these children will be included into the piloting phase.

Recruitment In total, 20 children - 10 children with CP-A and 10 who are TD as healthy controls - aged between 10 to 16 years old will be recruited. The children in the two groups will be matched for age, BMI, and physical activity level.

Study 1: Addressing aim 1-2 - Development of an exercise-application Methodology: Workshops to further develop the eHealth app: Four separate workshops will then be conducted to discuss the functions and the setup of communication of the initial prototype, as well as how to deliver the exercise sessions and what they preferably may contain. Workshop 1 will consist of 4-6 children children with CP-A and TD. Workshop 2 will consist of family caregivers. Workshop 3 of professional caregivers as physiotherapists and workshop 4 of sport professionals as personal trainers. The workshops will employ a participatory approach, enabling active contributions from participants and be facilitated by researchers from the research group. After the workshops, the eHealth app will be updated by a technician based on the feedback received.

Study 2: Addressing aim 3 - Feasibility testing of an exercise-application Methodology: Four children in each group, in total eight children, will take part in the feasibility analysis. During the first three weeks will the children be supervised at schedule timepoints through an eHealth solution and during the last three weeks the children follows pre-recorded exercise sessions at a suitable time for the family.

After the first 6 weeks of exercise training procedural, clinical and methodological uncreates will be analysed. Feedback from the participants and their family-caregivers, will be collected through semi-structured interviews to evaluate the feasibility of the exercise training intervention. Depending on the findings during the feasibility testing, the exercise training intervention may change.

DATA ANALYS AND STATISTIC A mixed method approach will be used to meet the aims of the project and collect both quantitative and qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* children with CP-A defined as GMFCS-E&R I-II
* children who are TD and not participating in any regular and planned leisure time physical exercise will be included in the study.

Exclusion Criteria:

* Ambulant children with CP walking with a walking aid (GMFCS-E&R III);
* ambulant children who are TD with other neurological diagnoses, metabolic diagnoses, orthopaedic disabilities, asthma, heart diseases, cognitive impairment, or indigestion of regular medication.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Complaiance to the exercise regim | From the start of exercise period 1 to the end of exercise period 2 in total 20 weeks.
  Number of exercise sessions performed

SECONDARY OUTCOMES:
Variance in the predefinde workload | From the start of exercise period 1 to the end of exercise period 2 in total 20 weeks.
  Coefficient of variance during each exercise session assessed by the spinning bike.
Number of adversed events due to illness | From the start of exercise period 1 to the end of exercise period 2 in total 20 weeks.
  Number registered in the ehealth app
Number of adverse avents due to technical issues | From the start of exercise period 1 to the end of exercise period 2 in total 20 weeks.
  Number registered in the ehealth app
Maximal exercise capacity | From inclusion in the study undtil the last exercise test in total 20 weeks.
  Indirect calorimetry will be used during a maximal incremental exercise test. The exercise test will be initiated by cycling on a cycle ergometer for 6 minutes at 30 W, followed by an increase of 10W/minute until exhaustion. The test will performed before and after each exercise period.
  Exercise tests will be performed on a cycle ergometer (Monark 936, Monark Exercise AB, Vansbro, Sweden). An airtight mask covering the mouth and nose will be worn to measure breath-by-breath of VO2 and VCO2, for determination of maximal oxygen consumption (VO2peak), maximal workload (WRpeak), oxygen kinetics and Respiratory Exchange Ratio (RER) (Oxycon Mobile, Jaeger, Germany). Heart rate will be recorded continuously throughout the test (Polar, Finland).

OTHER OUTCOMES:
Experiance | From inclusion in the study until the last exercise test in total 20 weeks.
  Semi-structured interviews
Usability | From inclusion in the study until the last exercise test in total 20 weeks.
  Usability questinnary

CONTACTS AND LOCATIONS:
Overall Officials: Åsa B Tornberg, Associate Professor, Principal Investigator — Department of Health Sciences, Medical Faculty, Lund Univeristy, Sweden
Locations (1):
- Medical Faculty, Lund University, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
A small study group with risk of identification of individuals